CLINICAL TRIAL: NCT06623240
Title: A Randomized, Double-Blind, Phase 2, Efficacy and Safety Cross-Over Study of Allogeneic HB-adMSCs vs Placebo for the Treatment of Oligoarticular and Polyarticular Juvenile Idiopathic Arthritis
Brief Title: HB-adMSCs vs Placebo for the Treatment of Juvenile Idiopathic Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In the time that the site has been active, there have been 0 patients enrolled despite our best efforts. It is clear that it is not feasible to conduct this study at this time; therefore, we have withdrawn this study.
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBJIA01
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: JIA; juvenile idiopathic arthritis; juvenile arthritis; oligoarticular; polyarticular; polyarticular juvenile idiopathic arthritis; oligoarticular juvenile idiopathic arthritis; arthritis
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, Phase 2, efficacy and safety cross-over study of allogeneic HB-adMSCs vs placebo for the treatment of oligoarticular and polyarticular juvenile idiopathic arthritis. Cohort 1 (first 6 patients) will undergo a screening period (up to 35 days) and an 8-week active treatment period, followed by a 64-week follow-up. Cohort 2 (remaining 60 patients) will undergo a screening period (up to 35 days), an 8-week active treatment period and an 8-week inactive treatment period (placebo) with a washout period of 12 weeks between the treatment periods. Subjects assigned to Cohort 2 - Group AB will receive allogeneic HB-adMSCs before the washout period, while subjects assigned to Cohort 2 - Group BA will receive allogeneic HB-adMSCs after the washout period. Group AB will undergo a safety follow-up of 64 weeks after their last infusion of HB-adMSCs, while Group BA will undergo a safety follow-up of 44 weeks after their last infusion of HB-adMSCs.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This clinical trial is a double-blinded study, meaning that the subjects and the researchers both do not know the group assignments. Research staff and subjects may be unblinded once all study data has been collected, all study-related procedures and follow-ups are completed, and all monitoring has been completed. (The first 6 patients (Cohort 1) will only receive active treatment; therefore, blinding is not applicable).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 2: Group AB (Experimental): Cohort 2 - Group AB will receive allogeneic HB-adMSCs (Hope Biosciences adipose-derived mesenchymal stem cells) at study weeks 0, 4, and 8. Then, Group AB will receive placebo (Sterile Saline Solution 0.9%) at weeks 20, 24, and 28 after a washout period of 12 weeks between active treatment and placebo.
  Interventions: Biological: allogeneic Hope Biosciences adipose-derived mesenchymal stem cells; Other: Normal Saline Solution 0.9%
- Cohort 2: Group BA (Experimental): Cohort 2 - Group BA will receive placebo (Sterile Saline Solution 0.9%) at study weeks 0, 4, and 8. Then, Group BA will receive allogeneic HB-adMSCs (Hope Biosciences adipose-derived mesenchymal stem cells) at weeks 20, 24, and 28 after a washout period of 12 weeks between placebo and active treatment.
  Interventions: Biological: allogeneic Hope Biosciences adipose-derived mesenchymal stem cells; Other: Normal Saline Solution 0.9%
- Cohort 1: Group A (Experimental): Cohort 1 - Group A will receive allogeneic HB-adMSCs (Hope Biosciences adipose-derived mesenchymal stem cells) at study weeks 0, 4, and 8.
  Interventions: Biological: allogeneic Hope Biosciences adipose-derived mesenchymal stem cells

INTERVENTIONS:
Biological: allogeneic Hope Biosciences adipose-derived mesenchymal stem cells — Product: Allogeneic HB-adMSCs (Hope Biosciences adipose derived mesenchymal stem cells)
  Dose determined by body weight:
  * 50 million cells in 50mL saline: ≥ 10 kg to < 22 kg
  * 100 million cells in 100mL saline: ≥ 22 kg to < 45 kg
  * 200 million cells in 250mL saline: ≥ 45 kg Route: Intravenous Regimen: Weeks 0, 4, and 8 (Cohort 1: Group A and Cohort 2: Group AB) or Weeks 20, 24, and 28 (Cohort 2: Group BA)
Other: Normal Saline Solution 0.9% — Product: Normal Saline Solution 0.9% Route: Intravenous Regimen: Weeks 0, 4, and 8 (Cohort 2: Group BA) or Weeks 20, 24, and 28 (Cohort 2: Group AB)
  Arms: Cohort 2: Group AB; Cohort 2: Group BA

SUMMARY:
Methodology: Randomized, double-blind, AB/BA cross-over study with a washout period of 12 weeks.

Treatment Duration: 8 weeks per group

General Objectives: To assess the efficacy and safety of multiple intravenous infusions of allogeneic HB-adMSCs by improving signs and symptoms of juvenile idiopathic arthritis in this subject population.

Number of Subjects: 66 (6 subjects in Cohort 1 and 60 subjects in Cohort 2)

Indication: Juvenile Idiopathic Arthritis

DETAILED DESCRIPTION:
Primary Objectives:

* To assess the safety of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with oligoarticular or polyarticular juvenile idiopathic arthritis as determined by the incidence of adverse events or serious adverse events. (Time Frame: Week 0 to Week 72).
* To investigate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with oligoarticular or polyarticular juvenile idiopathic arthritis as determined by improvements in ACR Pedi 30 scores. (Time Frame: Week 0 to Week 52 for Group AB and Week 0 to Week 72 for Group BA).

Secondary Objectives

* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with oligoarticular or polyarticular juvenile idiopathic arthritis as determined by improvements in ACR Pedi 50 scores. (Time Frame: Week 0 to Week 52 for Group AB and Week 0 to Week 72 for Group BA).
* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with oligoarticular or polyarticular juvenile idiopathic arthritis as determined by improvements in ACR Pedi 70 scores. (Time Frame: Week 0 to Week 52 for Group AB and Week 0 to Week 72 for Group BA).
* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with oligoarticular or polyarticular juvenile idiopathic arthritis as determined by improvements in CRP values. (Time Frame: Week 0 to Week 52 for Group AB and Week 0 to Week 72 for Group BA).
* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with oligoarticular or polyarticular juvenile idiopathic arthritis as determined by improvements in ESR values. (Time Frame: Week 0 to Week 52 for Group AB and Week 0 to Week 72 for Group BA).
* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with oligoarticular or polyarticular juvenile idiopathic arthritis as determined by improvements in Peds QL scores. (Time Frame: Week 0 to Week 52 for Group AB and Week 0 to Week 72 for Group BA).

ELIGIBILITY:
Inclusion Criteria:

The subject will be eligible for inclusion in this clinical trial only if all of the following criteria apply:

1. Male and female subjects who are ≥ 2 years old and < 17 years old.

   a.The first 6 subjects enrolled must be ≥ 12 years old and < 17 years old
2. Must be diagnosed with Oligoarticular or Polyarticular Juvenile Idiopathic Arthritis by a Pediatric Rheumatologist.
3. Must have rheumatoid factor (RF) factor test result documented in medical records.
4. Must have at least 3 affected joints at the screening visit.
5. Must have a body weight of > 10 kg at the screening visit.
6. Subjects without a current established treatment for JIA who are not on treatment because they have failed at least 2 approved medications for their condition, or if being treated, subjects who are on a stable dose of arthritis therapy regimen for ≥3 months prior to screening.
7. Must have an abnormal CRP result and/or abnormal ESR result at screening. Abnormal C-reactive protein (CRP) value defined as > 1 mg/dL. Abnormal Erythrocyte Sedimentation Rate (ESR) value defined as >15 mm/hr for males and >20 mm/hr for females.
8. Female study subjects of childbearing potential should not be pregnant or plan to become pregnant during study participation and for 6 months after the last investigational product administration. Female study subjects of childbearing potential must confirm usage of one of the following contraceptive measures:

   * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   * Barrier contraceptive methods (condoms, diaphragm, etc.).
9. Male subjects if their sexual partners can become pregnant should ensure the use one of the following methods of contraception during study participation and for 6 months after the last administration of the investigated product.

   * Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   * Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   * Barrier contraceptive methods (condoms, diaphragm, etc.).
10. Study subject's parent(s)/LAR is/are able and willing to comply with the requirements of this clinical trial.
11. Voluntarily signed informed consent from study subjects' parent(s) or legally authorized representative obtained before any clinical-trial related procedures are performed.

Exclusion Criteria:

The subject will not be eligible for inclusion in this clinical trial if any of the following criteria apply:

1. Study subject has any of the following laboratory results at the screening visit:

   1. WBC: <3000 cells/μL OR >15000 cells/μL (<3 K cells/μL or >15 K cells/μL)
   2. Hemoglobin: <8 g/dL
   3. Absolute Neutrophil Count: <1500 cells/μL
   4. Platelet: <150000 cells/μL (<150 K cells/μL)
   5. Sodium: <120 mEq/L OR >150 mEq/L
   6. Glucose: >150 mg/dL
   7. Potassium: <3.5 mEq/L OR >6 mEq/L
   8. BUN: >25 mg/dL
   9. Creatinine: >2 mg/dL
   10. BUN/Creatinine ratio: >50
   11. AST: >100 U/L
   12. ALT: >100 U/L
2. Study participant has any vital sign abnormalities at the screening visit as determined by the investigator.
3. Study subject has 1 or more significant uncontrolled concurrent medical conditions (verified by medical records), including the following:

   1. Diabetes Mellitus
   2. Crohn's Disease
   3. Lupus
   4. Multiple Sclerosis
4. Study subject has any active malignancy, including evidence of cutaneous basal, squamous cell carcinoma or melanoma.
5. Study subject has known alcoholic addiction or dependency or has current substance use or abuse.
6. Study subject has received any stem cell treatment within 1 year before first dose of investigational product other than stem cells produced by Hope Biosciences LLC.
7. Receiving any investigational therapy or any approved therapy for investigational use within 1 year prior first dose of the investigational product other than COVID-19 vaccines.
8. Study subject has any other laboratory abnormality or medical condition which, in the opinion of the investigator, poses a safety risk or will prevent the subject from completing the study.
9. Study subject's parent(s)/LAR unable to understand and provide signed informed consent.
10. Study subject and/or study subject's parent(s)/LAR unlikely to complete the study or adhere to the study procedures.
11. Study subject with known concurrent acute or chronic viral hepatis B or C or human immunodeficiency virus (HIV) infection.
12. Study subject with any systemic infection requiring treatment with antibiotics, antivirals, or antifungals within 30 days prior to first dose of the investigational product.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs). | Baseline (Week 0) up to Week 72
  Treatment-emergent adverse events are defined as any adverse events which occur after the first infusion with HB-adMSCs up to the week 12 visit for Group AB or the week 32 visit for group BA.
Incidence of serious adverse events (SAEs). | Baseline (Week 0) up to Week 72
  Incidence of serious Adverse Events (SAEs)
Incidence and risk of AEs of particular interest (serious or nonserious) | Baseline (Week 0) up to Week 72
  Incidence and risk of AEs of particular interest (serious or nonserious), including thromboembolic events, infections, and hypersensitivities.
Changes from Baseline in laboratory values results - Complete Blood Count (x10^3 Cells/uL) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (x10^3 Cells/uL)
Changes from Baseline in laboratory values results - Complete Blood Count (% of WBC) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (% of WBC)
Changes from Baseline in laboratory values results - Complete Blood Count (pg) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (pg)
Changes from Baseline in laboratory values results - Complete Blood Count (g/dL) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (g/dL)
Changes from Baseline in laboratory values results - Complete Blood Count (fL) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (fL)
Changes from Baseline in laboratory values results - Complete Blood Count (x10^6 Cells/uL) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (x10^6 Cells/uL)
Changes from Baseline in laboratory values results - Complete Blood Count (% Difference in Volume and Size of RBC) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (% Difference in Volume and Size of RBC)
Changes from Baseline in laboratory values results - Complete Blood Count (% of Total Blood Cell Count) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (% of Total Blood Cell Count)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (g/dL) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (g/dL)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Albumin to Calc. Globulin) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Albumin to Calc. Globulin)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (U/L) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (U/L)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mg/dL) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mg/dL)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mEq/L) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mEq/L)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mL/Min/1.73m^2) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mL/Min/1.73m^2)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Calc BUN/Creatinine) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Calc BUN/Creatinine)
Changes from Baseline in laboratory values results - Coagulation Panel (Seconds) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Coagulation Panel (Seconds)
Changes from Baseline in laboratory values results - Coagulation Panel (Ratio of Prothrombin Time/Mean Prothrombin Time) | Baseline (Week 0) up to Week 72
  Clinically significant changes from Baseline in laboratory values results - Coagulation Panel (Ratio of Prothrombin Time/Mean Prothrombin Time)
Changes from Baseline in Vital Signs - Respiratory Rate (Breaths per minute) | Baseline (Week 0) up to Week 72
  Clinically significant changes from baseline in Respiratory Rate (Breaths per minute)
Changes from Baseline in Vital Signs - Heart Rate (Breaths per minute) | Baseline (Week 0) up to Week 72
  Clinically significant changes from baseline in Heart Rate (Breaths per minute)
Changes from Baseline in Vital Signs - Body Temperature (Celsius) | Baseline (Week 0) up to Week 72
  Clinically significant changes from baseline in Body Temperature (Celsius)
Changes from Baseline in Vital Signs - Systolic Blood Pressure (mmHg) | Baseline (Week 0) up to Week 72
  Clinically significant changes from baseline in Systolic Blood Pressure (mmHg)
Changes from Baseline in Vital Signs - Diastolic Blood Pressure (mmHg) | Baseline (Week 0) up to Week 72
  Clinically significant changes from baseline in Diastolic Blood Pressure (mmHg)
Changes from Baseline in Vital Signs - SPO2 (%) | Baseline (Week 0) up to Week 72
  Clinically significant changes from baseline in SPO2 (%)
Clinically significant changes in weight results (in kg) | Baseline (Week 0) up to Week 72
  Changes from Baseline in weight results in patients (in kg)
Number of participants with abnormal physical examination results - Abdomen | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Abdomen
Number of participants with abnormal physical examination results - Cardiovascular | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Cardiovascular
Number of participants with abnormal physical examination results - Head, Eyes, Ears, Nose, and Throat | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Head, Eyes, Ears, Nose, and Throat
Number of participants with abnormal physical examination results - Lymph Node | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Lymph Node
Number of participants with abnormal physical examination results - Musculoskeletal | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Musculoskeletal
Number of participants with abnormal physical examination results - Neurological | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Neurological
Number of participants with abnormal physical examination results - Respiratory | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Respiratory
Number of participants with abnormal physical examination results - Skin | Baseline (Week 0) up to Week 72
  Number of participants with abnormal physical examination results - Skin
Clinically significant changes in ACR Pedi 30 | Baseline (Week 0) up to Week 52 for Group AB or Week 72 for Group BA
  Changes from Baseline in ACR Pedi 30 in patients

SECONDARY OUTCOMES:
Clinically significant changes in ACR Pedi 50 | Baseline (Week 0) up to Week 52 for Group AB or Week 72 for Group BA
  Changes from Baseline in ACR Pedi 50 in patients
Clinically significant changes in ACR Pedi 70 | Baseline (Week 0) up to Week 52 for Group AB or Week 72 for Group BA
  Changes from Baseline in ACR Pedi 70 in patients
Clinically significant changes in C-reactive protein values (mg/L) | Baseline (Week 0) up to Week 52 for Group AB or Week 72 for Group BA
  Changes from Baseline in C-reactive protein values in patients (mg/L)
Clinically significant changes in erythrocyte sedimentation rate values (mm/h) | Baseline (Week 0) up to Week 52 for Group AB or Week 72 for Group BA
  Changes from Baseline in erythrocyte sedimentation rate values in patients (mm/h)
Clinically significant changes in PedsQL | Baseline (Week 0) up to Week 52 for Group AB or Week 72 for Group BA
  Changes from Baseline in PedsQL in patients

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Research Foundation
Locations (1):
- Hope Biosciences Research Foundation, Sugar Land, Texas, United States